CLINICAL TRIAL: NCT06033235
Title: Impact of Computed Tomography Scanning on ICU Patient Management: Retrospective Study
Brief Title: Computed Tomography Scanning in ICU
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Other Study IDs: 0220-23-MMC
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: CT Scans in the Intensive Care Unit
MeSH Terms: interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CT scan in critically ill patients in the intensive care unit — CT scan in critically ill patients in the intensive care unit

SUMMARY:
Patients admitted to the intensive care unit often require CT imaging. Performing this diagnostic test on a critically ill patient involves risks, such as those associated with transferring a ventilated and unstable patient and those associated with the injection of intravenous contrast material. Also, multiple CT examinations may create a burden on the X-ray institute and the medical staff, result in the postponement of CT examinations for other patients, as well as increase hospitalization costs.

In this work, we would like to check the rate of complications involved in performing a CT scan in patients hospitalized in the general intensive care unit of our institution, while analyzing the differences between the times the test is performed (morning, night shift), as well as examine in what percentage of the CT scans the test performed contributed to a significant progress in the diagnosis or a significant change in the treatment plan of the patient, while referring to subgroups (sepsis, trauma, respiratory failure, with an emphasis on covid patients, patients with scoliosis, patients with intracranial pathology).

ELIGIBILITY:
Inclusion Criteria:All patients who underwent CT examinations during hospitalization in the intensive care unit for any etiology, from January 2020 to January 2023.

-

Exclusion Criteria:Patients who did not meet the above criteria or for whom data were missing.

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent CT examinations during hospitalization in the intensive care unit for any etiology, from January 2020 to January 2023.
  -
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Change in diagnosis and/or patient management | 3 years
  To examine in what percentage of the CT examinations the examination contributed to a significant progress in the diagnosis or a significant change in the patient's treatment plan, while referring to subgroups of patients in the intensive care unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No